CLINICAL TRIAL: NCT06353438
Title: Implementation of a Community Based Exercise Program for Older Adults Using Hydraulic Resistance Equipment
Brief Title: Hydraulic Resistance and Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Staten Island, the City University of New York (Other)
Collaborators: Bay Ridge Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024XXXX
Record Dates: First submitted 2024-03-20; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Aging; Fall; Old Age; Debility; Muscle Weakness
MeSH Terms: conditions — Frailty; Muscle Weakness | interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All subjects will participate in a 2x/week for 6 weeks exercise program using Frei FACTUM® novus II line exercise equipment, which uses hydraulic resistance. Each session will take 30-45 minutes to complete. The equipment uses concentric movements only but works both agonist and antagonist muscles with each piece of equipment (IE: push and pull). Participants results will be compared pre and post intervention.
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Exercise Program — Concentric strengthening of multiple muscle groups 2x/week for 6 weeks.

SUMMARY:
The goal of this quasi-experimental study using a pre and post test design is to learn about the effect of participating in an exercise program with hydraulic exercise equipment on fall risk in the older adult population. The main questions it aims to answer are:

* Does the use of hydraulic exercise equipment decrease fall risk in older adults?
* Does the use of hydraulic exercise equipment improve function in older adults?

Participants will be evaluated pre and post intervention for strength, fall risk using Berg Balance Scale, Tinetti Balance and Gait Assessment, Timed Up and Go, and functional ability using the Lower Extremity Functional Scale. Participants will engage in an exercise program using 5 different pieces of hydraulic exercise equipment (Frei FACTUM® novus II line) 2x/week for for 6 weeks for 30-45 minutes each session. The equipment uses concentric movements only and works agonist and antagonist muscles with each machine (IE: push and pull, both concentric).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age 60+

Exclusion Criteria:

* Age <60
* Neurological condition
* Surgery within last 6 months
* Current injury
* Inability to follow directions
* Inability to participate in physical activity for any medical reason

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 1 week prior to intervention start date (pre-test) and 1 week post intervention end date (post-test)
  Objective functional outcome measure that assesses fall risk. Participants will move through 14 different tasks and will be assessed on their performance on a 0-4 scale. The higher the number given for a task, the better the participant's balance. The highest possible score is 56, which indicates low fall risk. The lower the score, the higher the fall risk. Minimal detectable change ranges from 5-7 depending on the diagnosis of the patient.
Timed Up and Go | 1 week prior to 1 week prior to intervention start date (pre-test) and 1 week post intervention end date (post-test) start date and 1 week post intervention end date
  Objective functional outcome measure that assesses fall risk. Participants will start seated in a chair. When the assessor says "Go" the participant will stand up from the chair, walk 3 meters or 10 feet, turn around and walk back to the chair and sit down. The assessor will use a stopwatch to measure how much time it takes to complete this task. A score of 12 seconds or more indicates increased fall risk.
Tinetti Balance and Gait Assessment Tool | 1 week prior to intervention start date (pre-test) and 1 week post intervention end date (post-test)
  Objective functional outcome measure that assesses fall risk. This test looks at 9 different balance tasks (sitting balance, sit to stand, standing balance, for example) and 7 domains during gait (hesitancy to begin walking, step length and height, step symmetry, step continuity, for example). Balance score is out of 16 and gait score is out of 12. Total score is out of 28. The lower the score, the higher the fall risk.
Lower Extremity Functional Scale | 1 week prior to intervention start date (pre-test) and 1 week post intervention end date (post-test)
  Objective functional outcome measure that determines functional ability during lower extremity tasks. Subjects rate their ability to perform 20 different lower extremity tasks on a 0-4 scale (0 is unable to complete activity and 4 is no difficulty). Scores range from 0-80. A total score of 80 means no difficulty with any task listed. 0 means unable to perform any task listed. The minimum clinically important difference (MCID) for the Lower Extremity Functional Scale is 9 points.

SECONDARY OUTCOMES:
Strength | 1 week prior to intervention start date and 1 week post intervention end date
  Participant strength will be measured using the exercise equipment (FREI-Swiss Factum Line). Participants will perform maximal voluntary isometric contractions (MVIC) for each muscle group on each piece of exercise equipment for agonist and antagonist muscles. This strength testing will determine how much resistance will be provided during the intervention; the exercise equipment uses a specific algorithm to determine how much load will be provided. Each participant will be given a unique card to "log in" to the equipment during each session and it will keep note of their scores and performance on each piece of equipment. The MVIC will take place pre and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda L Rotondo, DPT, Principal Investigator — CUNY College of Staten Island
Locations (1):
- Bay Ridge Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
There will be 1 PI and 5 co-investigators for this study. Data will be shared with those involved for data analysis purposes. Data will be stored in the PI's locked office in a locked filing cabinet and on a password protected computer owned by the PI.